CLINICAL TRIAL: NCT02324010
Title: Effects of Sitagliptin on Postprandial Glycaemia, Incretin Hormones and Blood Pressure in Type 2 Diabetes - Relationship to Gastric Emptying
Brief Title: Effects of Sitagliptin on Gastric Emptying, Glycaemia and Blood Pressure in Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Adelaide Hospital (Other)
Responsible Party: Principal Investigator, Karen Jones, Professor, Royal Adelaide Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 140916
Record Dates: First submitted 2014-12-16; First posted 2014-12-24 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Gastroparesis; Diabetes Mellitus
Keywords: gastric emptying; glycemia; appetite; incretin hormones
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus | interventions — Sitagliptin Phosphate; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitaglipltin (100mg) (Experimental): Active drug (sitagliptin)
  Interventions: Drug: Placebo
- Placebo (sugar pill) (Placebo Comparator): Inactive drug (placebo)
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — 100mg mane for 2 days
  Other Names: MK-0431-075, Januvia
  Arms: Placebo (sugar pill)
Drug: Placebo — Inactive drug (Placebo)
  Other Names: Sugar pill
  Arms: Sitaglipltin (100mg)

SUMMARY:
The purpose of this study is to evaluate the acute effects of sitagliptin on postprandial glycemia, incretin hormones and blood pressure, and the relationship to gastric emptying, after a mashed potato meal in patients with type 2 diabetes.

DETAILED DESCRIPTION:
The purpose of this study is to (i) evaluate the acute effects of the dipeptidyl peptidase-4 (DPP-4) inhibitor, sitagliptin (100mg once daily for two days), on gastric emptying, postprandial plasma glucose, insulin, glucagon and 'incretin' hormones (ie. glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP)), blood pressure and heart rate after a high carbohydrate meal, and (ii) to determine whether the magnitude of the effects of sitagliptin on postprandial glycaemia and blood pressure is related to the rate of gastric emptying, in patients with type 2 diabetes.

The rate of entry of carbohydrate into the small intestine is especially important in patients with diabetes mellitus. Sitagliptin is an orally administered inhibitor of dipeptidyl-peptidase-IV (DPP-IV), the enzyme responsible for the degradation of GLP-1. It is hypothesized that sitagliptin will increase the GLP-1 response to, and thereby slow gastric emptying and diminish the glycaemic and blood pressure response to, a carbohydrate-containing meal.

Twenty healthy subjects (male and female) will be studied. Each subject will be studied on two occasions following treatment for 2 days with sitagliptin (100mg once daily) or matching placebo in a randomized, double blind, crossover design. Measurements of gastric emptying, intragastric meal distribution, blood glucose concentrations, gut hormones, blood pressure, splanchnic flow and appetite will be measured for 4 hours following ingestion of a mashed potato meal.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (World Health Organisation (WHO) criteria), managed by diet or metformin alone
* Body mass index (BMI) 20 - 40 kg/m2
* Males and females (females of reproductive potential must be using an appropriate contraceptive method)
* Glycated haemoglobin (HbA1c) ≤ 8.5%
* Haemoglobin above the lower limit of the normal range (i.e. >135g/L for men and 115g/L for women), and ferritin above the lower limit of normal (i.e. >10mcg/L)

Exclusion Criteria:

* Subjects with gastrointestinal disease, significant upper or lower gastrointestinal symptoms, or previous gastrointestinal surgery (other than uncomplicated appendicectomy or cholecystectomy)
* Other significant illness, including epilepsy, cardiovascular or respiratory disease.
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy.
* Impaired renal or liver function (as assessed by calculated creatinine clearance < 50 mL/min using the Cockroft-Gault equation (27) or abnormal liver function tests (> 2 times upper limit of normal range)).
* Requirement for medication known to influence blood pressure and/or heart rate and/or gastrointestinal function, drugs with anticholinergic effects
* Alcohol consumption > 20 g per day
* Smoking > 10 cigarettes per day
* Pregnancy or lactation.
* Vegetarian
* Allergy to sitagliptin or any other 'gliptin'.
* Donation of blood within the previous 3 months
* Participation in any other research studies within the previous 3 months
* Exposure to ionising radiation for research purposes in the previous 12 months
* Inability to give informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Gastric emptying | 3 hours per gastric emptying study (i.e. 6 hours)
  Gastric retention (percent in the total stomach)

SECONDARY OUTCOMES:
Glycaemia | 4 hours during each gastric empty study (i.e. 8 hours)
  blood glucose (mmol/L) and plasma insulin (mU/L)
Gastrointestinal hormone release | 4 hours during each gastric empty study (i.e. 8 hours)
  GLP-1, GIP, C-peptide, 3-OMG
Intragastric meal distribution | 3 hours during each gastric empty study (i.e. 6 hours)
  percent retention in the proximal and distal stomach
Blood pressure | 4.5 hours during each gastric empty study (i.e. 9 hours)
  systolic and diastolic blood pressure (mmHg)
Heart rate | 4.5 hours during each gastric empty study (i.e. 9 hours)
  Heart rate (beats per minute)
Splanchnic blood flow | 4 hours during each gastric empty study (i.e. 8 hours)
  Doppler ultrasound of superior mesenteric artery flow (ml/min)
Cardiac output | 4 hours during each gastric empty study (i.e. 8 hours)
  Finapres (L)
Stroke volume | 4 hours during each gastric empty study (i.e. 8 hours)
  Finapres (mL)
Appetite | 4 hours during each gastric empty study (i.e. 8 hours)
  visual analogue questionnaire to assess hunger, fullness, desire to eat (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Jones, DAppSci, PhD, Principal Investigator — University of Adelaide
Locations (1):
- University of Adelaide, Discipline of Medicine, Royal Adelaide Hospital, Adelaide, South Australia, Australia

REFERENCES:
- [Background] Wu T, Rayner CK, Young RL, Horowitz M. Gut motility and enteroendocrine secretion. Curr Opin Pharmacol. 2013 Dec;13(6):928-34. doi: 10.1016/j.coph.2013.09.002. Epub 2013 Sep 20. PMID 24060702
- [Background] Chaikomin R, Rayner CK, Jones KL, Horowitz M. Upper gastrointestinal function and glycemic control in diabetes mellitus. World J Gastroenterol. 2006 Sep 21;12(35):5611-21. doi: 10.3748/wjg.v12.i35.5611. PMID 17007012
- [Background] Horowitz M, Edelbroek MA, Wishart JM, Straathof JW. Relationship between oral glucose tolerance and gastric emptying in normal healthy subjects. Diabetologia. 1993 Sep;36(9):857-62. doi: 10.1007/BF00400362. PMID 8405758
- [Background] Jones KL, Horowitz M, Carney BI, Wishart JM, Guha S, Green L. Gastric emptying in early noninsulin-dependent diabetes mellitus. J Nucl Med. 1996 Oct;37(10):1643-8. PMID 8862300
- [Background] Horowitz M, Rayner CK, Jones KL. Mechanisms and clinical efficacy of lixisenatide for the management of type 2 diabetes. Adv Ther. 2013 Feb;30(2):81-101. doi: 10.1007/s12325-013-0009-4. Epub 2013 Feb 13. PMID 23423907
- [Background] Baggio LL, Drucker DJ. Biology of incretins: GLP-1 and GIP. Gastroenterology. 2007 May;132(6):2131-57. doi: 10.1053/j.gastro.2007.03.054. PMID 17498508
- [Background] ELRICK H, STIMMLER L, HLAD CJ Jr, ARAI Y. PLASMA INSULIN RESPONSE TO ORAL AND INTRAVENOUS GLUCOSE ADMINISTRATION. J Clin Endocrinol Metab. 1964 Oct;24:1076-82. doi: 10.1210/jcem-24-10-1076. No abstract available. PMID 14228531
- [Background] Nauck M, Stockmann F, Ebert R, Creutzfeldt W. Reduced incretin effect in type 2 (non-insulin-dependent) diabetes. Diabetologia. 1986 Jan;29(1):46-52. doi: 10.1007/BF02427280. PMID 3514343
- [Background] Nauck MA, Heimesaat MM, Orskov C, Holst JJ, Ebert R, Creutzfeldt W. Preserved incretin activity of glucagon-like peptide 1 [7-36 amide] but not of synthetic human gastric inhibitory polypeptide in patients with type-2 diabetes mellitus. J Clin Invest. 1993 Jan;91(1):301-7. doi: 10.1172/JCI116186. PMID 8423228
- [Background] Nauck MA, Niedereichholz U, Ettler R, Holst JJ, Orskov C, Ritzel R, Schmiegel WH. Glucagon-like peptide 1 inhibition of gastric emptying outweighs its insulinotropic effects in healthy humans. Am J Physiol. 1997 Nov;273(5):E981-8. doi: 10.1152/ajpendo.1997.273.5.E981. PMID 9374685
- [Background] Khoo J, Rayner CK, Jones KL, Horowitz M. Incretin-based therapies: new treatments for type 2 diabetes in the new millennium. Ther Clin Risk Manag. 2009 Jun;5(3):683-98. doi: 10.2147/tcrm.s4975. Epub 2009 Aug 20. PMID 19707284
- [Background] Stevens JE, Horowitz M, Deacon CF, Nauck M, Rayner CK, Jones KL. The effects of sitagliptin on gastric emptying in healthy humans - a randomised, controlled study. Aliment Pharmacol Ther. 2012 Aug;36(4):379-90. doi: 10.1111/j.1365-2036.2012.05198.x. Epub 2012 Jun 28. PMID 22738299
- [Background] Vella A, Bock G, Giesler PD, Burton DB, Serra DB, Saylan ML, Dunning BE, Foley JE, Rizza RA, Camilleri M. Effects of dipeptidyl peptidase-4 inhibition on gastrointestinal function, meal appearance, and glucose metabolism in type 2 diabetes. Diabetes. 2007 May;56(5):1475-80. doi: 10.2337/db07-0136. Epub 2007 Feb 15. PMID 17303799
- [Background] Woerle H, Lindenberger T, Linke R, Foley JE, Ligueros-Sayalan AA, ZhangY, He Y-L, BelingerC, Goeke B, Schirra J. A single dose of vidagliptin (VILDA) decelerates gastric emptying (GE) in patients with type 2 diabetes (T2DM). American Diabetes Association, 67th Scientific Sessions 500-p (abstract), 2007.
- [Background] Wu T, Bound MJ, Zhao BR, Standfield SD, Bellon M, Jones KL, Horowitz M, Rayner CK. Effects of a D-xylose preload with or without sitagliptin on gastric emptying, glucagon-like peptide-1, and postprandial glycemia in type 2 diabetes. Diabetes Care. 2013 Jul;36(7):1913-8. doi: 10.2337/dc12-2294. Epub 2013 Jan 28. PMID 23359361
- [Background] Rayner CK, Samsom M, Jones KL, Horowitz M. Relationships of upper gastrointestinal motor and sensory function with glycemic control. Diabetes Care. 2001 Feb;24(2):371-81. doi: 10.2337/diacare.24.2.371. PMID 11213895
- [Background] Pilichiewicz AN, Chaikomin R, Brennan IM, Wishart JM, Rayner CK, Jones KL, Smout AJ, Horowitz M, Feinle-Bisset C. Load-dependent effects of duodenal glucose on glycemia, gastrointestinal hormones, antropyloroduodenal motility, and energy intake in healthy men. Am J Physiol Endocrinol Metab. 2007 Sep;293(3):E743-53. doi: 10.1152/ajpendo.00159.2007. Epub 2007 Jul 3. PMID 17609258
- [Background] Ma J, Pilichiewicz AN, Feinle-Bisset C, Wishart JM, Jones KL, Horowitz M, Rayner CK. Effects of variations in duodenal glucose load on glycaemic, insulin, and incretin responses in type 2 diabetes. Diabet Med. 2012 May;29(5):604-8. doi: 10.1111/j.1464-5491.2011.03496.x. PMID 22004512
- [Background] Jansen RW, Lipsitz LA. Postprandial hypotension: epidemiology, pathophysiology, and clinical management. Ann Intern Med. 1995 Feb 15;122(4):286-95. doi: 10.7326/0003-4819-122-4-199502150-00009. PMID 7825766
- [Background] Jones KL, Tonkin A, Horowitz M, Wishart JM, Carney BI, Guha S, Green L. Rate of gastric emptying is a determinant of postprandial hypotension in non-insulin-dependent diabetes mellitus. Clin Sci (Lond). 1998 Jan;94(1):65-70. doi: 10.1042/cs0940065. PMID 9505868
- [Background] Russo A, Stevens JE, Wilson T, Wells F, Tonkin A, Horowitz M, Jones KL. Guar attenuates fall in postprandial blood pressure and slows gastric emptying of oral glucose in type 2 diabetes. Dig Dis Sci. 2003 Jul;48(7):1221-9. doi: 10.1023/a:1024182403984. PMID 12870776
- [Background] Vanis L, Gentilcore D, Rayner CK, Wishart JM, Horowitz M, Feinle-Bisset C, Jones KL. Effects of small intestinal glucose load on blood pressure, splanchnic blood flow, glycemia, and GLP-1 release in healthy older subjects. Am J Physiol Regul Integr Comp Physiol. 2011 Jun;300(6):R1524-31. doi: 10.1152/ajpregu.00378.2010. Epub 2011 Mar 9. PMID 21389332
- [Background] Jian ZJ, Zhou BY. Efficacy and safety of acarbose in the treatment of elderly patients with postprandial hypotension. Chin Med J (Engl). 2008 Oct 20;121(20):2054-9. PMID 19080275
- [Background] Sasaki E, Goda K, Nagata K, Kitaoka H, Ohsawa N, Hanafusa T. Acarbose improved severe postprandial hypotension in a patient with diabetes mellitus. J Diabetes Complications. 2001 May-Jun;15(3):158-61. doi: 10.1016/s1056-8727(01)00138-6. PMID 11358685
- [Background] Gentilcore D, Bryant B, Wishart JM, Morris HA, Horowitz M, Jones KL. Acarbose attenuates the hypotensive response to sucrose and slows gastric emptying in the elderly. Am J Med. 2005 Nov;118(11):1289. doi: 10.1016/j.amjmed.2005.05.019. No abstract available. PMID 16271921
- [Background] Yonenaga A, Ota H, Honda M, Koshiyama D, Yagi T, Hanaoka Y, Yamamoto H, Yamaguchi Y, Iijima K, Akishita M, Ouchi Y. Marked improvement of elderly postprandial hypotension by dipeptidyl peptidase IV inhibitor. Geriatr Gerontol Int. 2013 Jan;13(1):227-9. doi: 10.1111/j.1447-0594.2012.00903.x. No abstract available. PMID 23286563
- [Background] Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. doi: 10.1159/000180580. PMID 1244564
- [Background] Trahair LG, Vanis L, Gentilcore D, Lange K, Rayner CK, Horowitz M, Jones KL. Effects of variations in duodenal glucose load on blood pressure, heart rate, superior mesenteric artery blood flow and plasma noradrenaline in healthy young and older subjects. Clin Sci (Lond). 2012 Mar;122(6):271-9. doi: 10.1042/CS20110270. PMID 21942924
- [Background] Parker BA, Sturm K, MacIntosh CG, Feinle C, Horowitz M, Chapman IM. Relation between food intake and visual analogue scale ratings of appetite and other sensations in healthy older and young subjects. Eur J Clin Nutr. 2004 Feb;58(2):212-8. doi: 10.1038/sj.ejcn.1601768. PMID 14749739
- [Background] Ahren B. DPP-4 inhibitors. Best Pract Res Clin Endocrinol Metab. 2007 Dec;21(4):517-33. doi: 10.1016/j.beem.2007.07.005. PMID 18054733
- [Background] Information JsP: Merck Sharp & Dohme (Australia) Pty Ltd. South Granville, NSW, Australia, 2008.
- [Background] Deacon CF. Dipeptidyl peptidase-4 inhibitors in the treatment of type 2 diabetes: a comparative review. Diabetes Obes Metab. 2011 Jan;13(1):7-18. doi: 10.1111/j.1463-1326.2010.01306.x. PMID 21114598